CLINICAL TRIAL: NCT02978417
Title: A Feasibility Study for Testing the Effects of Extended-release Naltrexone (Vivitrol) on Recidivism and Other Participant Outcomes in Drug Court Settings
Brief Title: Feasibility Study of Extended-release Naltrexone (Vivitrol) in Drug Court Settings
Acronym: DC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Laura and John Arnold Foundation (Other); Alkermes, Inc. (Industry); FHR (Fellowship Health Resources, Inc.) (Other); Wake County Recovery Court (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00074507; 69665 (Other Grant/Funding Number: Laura and John Arnold Foundation)
Record Dates: First submitted 2016-11-28; First posted 2016-12-01 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Opioid-Related Disorders
Keywords: Medication-assisted treatment; Drug Court; Pilot study; Opioid dependence; Criminal justice
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vivitrol (Active Comparator): All drug court clients in the pilot RCT will receive standard psychosocial treatment for opioid dependence from FHR as part of their drug court program participation. Participants randomized to Vivitrol® will receive standard treatment along with monthly Vivitrol® injections administered by study staff at outpatient visits. Vivitrol® is naltrexone for extended-release injectable suspension. It is an injectable suspension containing 380 mg of naltrexone in a microsphere formulation and 4 mL diluent. The recommended dose of Vivitrol® is 380 mg delivered intramuscularly every 4 weeks or once a month. The injection should be administered by a healthcare provider as an intramuscular (IM) gluteal injection, alternating buttocks for each subsequent injection (see Links section of PRS for more information about Vivitrol).
  Interventions: Drug: Naltrexone for extended-release injectable suspension
- Oral naltrexone (Active Comparator): Subjects randomized to oral naltrexone in addition to standard psychosocial treatment for opioid dependence from FHR as part of their drug court program participation. Oral naltrexone is the daily tablet formulation naltrexone that carries the same risks and benefits as the long-acting injectable formulation (Vivitrol®), except it does not have any of the risks related to injection (discomfort, potential for infection). Oral naltrexone is administered and provided by FHR to interested and eligible clients as part of the range of their usual care services.
  Interventions: Drug: Oral naltrexone

INTERVENTIONS:
Drug: Naltrexone for extended-release injectable suspension — Opioid-dependent Drug Court clients enrolled in the study will receive monthly injections of Vivitrol for up to 12 months if they continue to be medically eligible and willing.
  Other Names: Vivitrol
  Arms: Vivitrol
Drug: Oral naltrexone — Opioid-dependent Drug Court clients enrolled in the study will receive prescriptions for oral naltrexone for up to 12 months if they continue to be medically eligible and willing.
  Other Names: Revia
  Arms: Oral naltrexone

SUMMARY:
In preparation for a large-scale randomized controlled trial (RCT) of Vivitrol® effectiveness in drug courts, investigators propose a feasibility study in the Wake County, North Carolina drug court, where an estimated 50% of clients are opioid dependent.

Aim 1: Pilot RCT. Pilot-test the delivery of Vivitrol® treatment for 10-20 interested and eligible clients of the Wake County Drug Court.

DETAILED DESCRIPTION:
Aim 1. Pilot RCT. The pilot delivery of Vivitrol® in the Wake County Drug Court will be carried out with 20-40 eligible drug court clients under treatment by Fellowship Health Resources, Inc. (FHR), the community behavioral health treatment agency that is the contracted treatment provider for the Wake County Drug Court. Participants will be randomized in equal number to receive Vivitrol® plus treatment as usual (TAU) or TAU only. TAU for drug court clients receiving services at FHR includes psychosocial treatment such as individual or group therapy, and sometimes also oral naltrexone for clients who are medically eligible and interested in taking the medication, the cost of which is covered by the agency for uninsured clients. (FHR currently administers Vivitrol® for a small number of interested agency clients with health insurance that covers the medication; the vast majority of their drug court clients are uninsured and so have no real access to the extended-release formulation due to its high cost.) Vivitrol® is an FDA-approved extended-release injectable form of naltrexone. Naltrexone is also available in oral, but not extended release, form. Naltrexone is an opioid antagonist that "blocks" opioid receptors in the brain to stop pleasurable feelings associated with taking opioids. Potentially eligible subjects will be drug court-referred FHR clients willing and eligible to take Vivitrol®, and willing to be randomly assigned to Vivitrol® or TAU. Potential subjects already under treatment with oral naltrexone at FHR would be eligible to enter the study if willing to switch to injectable Vivitrol® if randomly assigned. Study subjects who are randomized to Vivitrol® would receive a once-monthly injection of Vivitrol® for 12 months, or less if they decide to stop receiving Vivitrol® or to drop out of the study. Those randomized to TAU would continue with treatment as before, which could including (1) staying on oral naltrexone if already on it, (2) considering starting oral naltrexone, if interested, or (3) continuing with psychosocial treatment only. The Vivitrol® will be administered by study medical personnel at FHR. Randomization to the Vivitrol® arm would add urine pregnancy testing to FHR's existing Vivitrol® medical evaluation protocol and consent process, which currently screens for pregnancy without requiring a urine test. A urine pregnancy test will be administered once per month for female study participants of child-bearing age who are in the Vivitrol® group. All drug court clients, including study participants in both study groups, have urine drug tests at least once per week as part of program participation.

In addition to participating in Vivitrol® and psychosocial treatment, pilot RCT participants will provide consent for FHR and the drug court to share information with the study team about their demographic and clinical characteristics, treatment participation (e.g., outpatient group therapy), and court-related events (e.g., type of conviction that led to their drug court participation, missed drug court appointments, sanctions for program violations, and the results of drug screens).

Participants will also provide two face-to-face interviews at baseline and 6 months after baseline, about their interest and experience in Vivitrol® and/or other medication-assisted treatment (MAT), other treatment preferences, level of functioning, quality of life, and engagement in employment or education.

Outcome measures include treatment participation, compliance with drug court conditions, arrests and incarcerations, treatment satisfaction, and self-reported subjective measures of functioning and quality of life.

If a participant chooses not to participate in the study at any time, it will not affect his/her relationship with the court, FHR, right to health care, or participation in the study interview data collection. Site staff will follow participants for the purposes of collecting research and safety information. Investigators discontinue Vivitrol® or oral naltrexone in circumstances such as: adverse reactions to the medication; a change in medical status that makes it unsafe for a participant to continue receiving the medication, including pregnancy; or a participant becoming ill during the study. Participants who discontinue Vivitrol® or oral naltrexone for any reason may continue to participate in interviews for the study.

ELIGIBILITY:
Inclusion Criteria:

* Client of Wake County Drug Treatment Court
* Interested in medication-assisted treatment for opioid dependence
* 18-65 years old
* understands and speaks English
* understands that study participation is fully voluntary, with no effect on court standing
* willing and able to give written informed consent
* has an opioid use disorder (DSM-5 diagnosis of moderate or severe opioid use disorder)
* has at least 6 months remaining before anticipated Drug Court graduation
* (if female) does not intend to become pregnant or breastfeeding during the study period and is willing to adhere to contraception requirements during the study period
* is willing to adhere to the study requirements
* Has at least 7-10 days without opioid use before beginning extended-release injectable naltrexone given that detoxification from opioids before initiating or resuming extended-release injectable naltrexone is necessary to prevent withdrawal.

Exclusion Criteria*:

* Is pregnant (i.e., has a positive pregnancy test), planning to become pregnant, or breastfeeding during the study
* Has a positive urine drug test for opioids, buprenorphine or methadone at the beginning of treatment and before each Vivitrol® injection
* Has used any opioid drug within 10 days prior to treatment
* Has a condition, disease state, previous medical history, or observed abnormalities (including physical examination, laboratory evaluation [e.g., kidney or liver function test result], or urinalysis finding) at screening that, in the opinion of the investigator, would preclude safe participation in the study or affect the ability of the subject to adhere to the protocol visit schedule, fulfill visit requirements, or would interfere with the study assessments, including, but not limited to, the following:

  * Uncontrolled hypertension, uncontrolled diabetes, renal disease/impairment, stroke, seizures or neurological disorder, cardiovascular (eg, endocarditis), neoplastic disease
  * Chronic pain condition requiring ongoing opioid analgesia
  * Aspartate aminotransferase or alanine aminotransferase value ≥3 times the upper limit of normal
  * Any contraindicated medical condition per the approved labeling for naltrexone
* Has had a DSM-5 diagnosis within the past 12 months of other psychiatric conditions or disorders that, in the investigator's opinion, could interfere with participation in the study
* Is currently physiologically dependent on any psychoactive substance (except caffeine, or tobacco) requiring medical intervention for detoxification
* Has a history of hypersensitivity or adverse reaction to naltrexone, or naloxone
* Has had significant suicidal ideation or behavior within the past year, as assessed with the Patient Health Questionnaire (PHQ-9)

  * Note about exclusion criteria: If, after joining the study, a subject has a positive drug test, becomes pregnant, or acquires another exclusion condition that would have prevented him/her from joining the study, he or she may remain in the study but will not be permitted to receive Vivitrol®. Study staff will continue to gather interview data and administrative data on any enrolled, willing subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison G Robertson, PhD, MPH, Principal Investigator — Department of Psychiatry & Behavioral Sciences, Duke University School of Medicine
Locations (1):
- Fellowship Health Resources (FHR), Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vivitrol prescribing information — http://www.Vivitrol.com/Content/pdf/prescribing_info.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community treatment provider Fellowship Health Resources (FHR) prescreened 19 people as eligible. Two declined to participate and 3 were terminated from court and lost eligibility, leaving 14 potential subjects.
Pre-assignment Details: Fourteen subjects consented to be in the study and completed a baseline interview. Four were terminated from court thereby losing eligibility, so they were not randomized.
Groups:
- Vivitrol: All drug court clients in the pilot RCT will receive standard psychosocial treatment for opioid dependence from FHR as part of their drug court program participation. Participants randomized to Vivitrol® will receive standard treatment along with monthly Vivitrol® injections administered by study staff at outpatient visits. Vivitrol® is an extended-release injectable suspension containing 380 mg of naltrexone in a microsphere formulation and 4 mL diluent. The recommended dose of Vivitrol® is 380 mg delivered intramuscularly every 4 weeks or once a month. The injection should be administered by a healthcare provider as an intramuscular (IM) gluteal injection, alternating buttocks for each subsequent injection (see Links section of PRS for more information about Vivitrol).
  Naltrexone for extended-release injectable suspension: Opioid-dependent Drug Court clients enrolled in the study will receive monthly injections of Vivitrol for up to 12
Period: Overall Study
Arm/Group | Vivitrol | Oral Naltrexone
Started | 5 | 5
Completed | 3 | 3
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vivitrol | Oral Naltrexone | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.4) | 37.4 (13.4) | 36.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Arrests
Description: Any new arrests during the 12-month study period. This information will be collected from administrative records.
Time Frame: 12 months
Population: Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 5 | 5
Participants | 2 | 2

2. Primary Outcome: Number of Participants With New Incarcerations
Description: Any new incarceration during the 12-month study period. This information will be collected from administrative records.
Time Frame: 12 months
Population: Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 5 | 5
Participants | 1 | 0

3. Secondary Outcome: Number of Positive Drug Screens
Description: Number of times a client had a positive drug screen. This information will be collected from administrative records.
Time Frame: 12 months
Population: Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Mean (Standard Deviation); unit: positive drug screens
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 5 | 5
positive drug screens | 2 (1.87) | 2.8 (2.59)

4. Secondary Outcome: Number of Sanctions Imposed by the Court
Description: Number of sanctions imposed by the court (e.g., brief stays in jail). This information will be collected from administrative records.
Time Frame: 12 months
Population: Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Mean (Standard Deviation); unit: sanctions
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 5 | 5
sanctions | 1.8 (1.30) | 3.6 (3.91)

5. Secondary Outcome: Number of Missed Court Appointments
Description: Number of missed court appointments during the 12-month study period. This information will be collected from administrative records.
Time Frame: 12 months
Population: Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Mean (Standard Deviation); unit: missed court appointments
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 5 | 5
missed court appointments | 0 (0) | 0 (0)

6. Secondary Outcome: Vivitrol Participation
Description: Number of Vivitrol injections from either arm of study. This information will be collected from administrative records.
Time Frame: 12 months
Population: Some subjects in the oral naltrexone arm received Vivitrol through other means. Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Mean (Standard Deviation); unit: Vivitrol injections
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 5 | 5
Vivitrol injections | 3.8 (4.97) | 1.4 (1.67)

7. Secondary Outcome: Treatment Participation (Non-Vivitrol)
Description: Number of oral naltrexone monthly prescriptions from either arm of study. This information will be collected from administrative records.
Time Frame: 12 months
Population: Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Mean (Standard Deviation); unit: oral naltrexone monthly prescriptions
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 5 | 5
oral naltrexone monthly prescriptions | 0.2 (0.45) | 1.6 (2.61)

8. Secondary Outcome: Change in Subjective Functioning: Medical Status
Description: Subjective assessment of medical status using the Addiction Severity Index (ASI) Lite (a single measure with multiple domains) collected via interviews at baseline and approximately six months.
Time Frame: Baseline, 6 months
Population: Data not collected.
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Who Reported Improvement in Subjective Functioning: Employment/Support Status
Description: Subjective assessment of employment opportunities collected via interviews at baseline and approximately six months.
Time Frame: Baseline, 6 months
Population: Subjects who completed the 6-month assessment. Due to the nature of this pilot phase study, all statistical analyses are considered exploratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 3 | 3
Participants | 1 | 2

10. Secondary Outcome: Number of Participants Who Reported Improvement in Substance Use
Description: Subjective assessment of alcohol/drug use in past 30 days collected via interviews at baseline and approximately six months.
Time Frame: Baseline, 6 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 3 | 3
Participants | 3 | 1

11. Secondary Outcome: Number of Participants Who Reported Illegal Behavior
Description: Subjective assessment of illegal behavior using the question, "Have you done anything that was against the law in the last 30 days?" collected via interviews approximately six months after baseline.
Time Frame: approximately 6 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

12. Secondary Outcome: Number of Participants Who Reported Improvement in Subjective Functioning: Family/Social Relationships
Description: Subjective assessment of family and social relationships using a single question about satisfaction with relationships over the past 30 days collected via interviews at baseline and approximately six months.
Time Frame: Baseline, approximately 6 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 3 | 3
Participants | 0 | 1

13. Secondary Outcome: Change in Subjective Functioning: Psychiatric Status
Description: Subjective assessment of psychiatric status using the Addiction Severity Index (ASI) Lite (a single measure with multiple domains) collected via interviews at baseline and approximately six months.
Time Frame: Baseline, approximately 6 months
Population: Data not collected.
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Treatment Satisfaction Score
Description: Reported as average of 12-item treatment satisfaction score at approximately six months. A score of 5 indicates strong agreement with positive statements about treatment satisfaction; a score of 0 indicates strong disagreement.
Time Frame: Approximately 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 3 | 3
score on a scale | 4.53 (0.75) | 4.83 (0.29)

15. Secondary Outcome: Change in Medication-assisted Treatment (MAT) Attitudes
Description: Change in MAT attitudes from baseline to follow-up. The average score of 4 questions about MAT for substance use disorder were calculated at baseline and follow-up, and the average score at baseline was subtracted from the average score at follow-up. The averages are based on questions for which a score of 5 indicates strong agreement with statements about MAT; a score of 1 indicates strong disagreement with such statements.
Time Frame: Baseline, approximately 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vivitrol | Oral Naltrexone
Number analyzed (Participants) | 3 | 3
score on a scale | 0.11 (0.59) | 0.08 (0.14)

ADVERSE EVENTS:
Time Frame: Approximately 6 months.
Arm/Group | Vivitrol | Oral Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 2/5 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vivitrol (N=5) | Oral Naltrexone (N=5)
Drug overdose (unrelated) (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vivitrol (N=5) | Oral Naltrexone (N=5)
Incarceration >5 days (Social circumstances) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT02978417/Prot_001.pdf